CLINICAL TRIAL: NCT00729352
Title: Dependency of O3-Induced Lung Mucus Hypersecretion on NQO1
Brief Title: Lung Mucus Hypersecretion and NQO1
Status: Completed | Type: Observational
Sponsor: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Responsible Party: Principal Investigator, Michael Foster, Professor, National Institute of Environmental Health Sciences (NIEHS)
Other Study IDs: 16347-CP-001; 00008404; R01ES016347 (NIH)
Record Dates: First submitted 2008-08-06; First posted 2008-08-07 (Estimated); Last update posted 2014-09-29 (Estimated); Status verified 2014-09

CONDITIONS: Environmental Exposure; Ozone; Air Pollution; Genetic Susceptibility
Keywords: NQO1, ozone, airway mucociliary clearance.
MeSH Terms: conditions — Genetic Predisposition to Disease

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Bronchoalveolar lavage specimens.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Control group: 18-35 yr old healthy subjects with wild type genotype for NQO1.
- Case group: 18-35 yr old healthy subjects who are homozygotic for minor allele of NQO1 Pro187Ser polymorphism

SUMMARY:
The research plan proposes translational studies in relevant animal models and human subjects in order to identify host (genetic) susceptibility factors that confer vulnerability to the prototypal air pollutant, ozone. The results will have significant impact upon, and aid in, understanding mechanisms regulating pro-oxidant lung injury, production and secretion of airway mucins, and clearance of respiratory mucus, and adverse health effects, that occur during and following exposure to airborne respiratory irritants.

DETAILED DESCRIPTION:
Recent epidemiologic studies have re-ignited an old controversy and opinions are forming as to whether mucus hypersecretion is crucial in the etiology of airway disease. For patients with asthma, chronic obstructive pulmonary disease (COPD), and cystic fibrosis, mucus hypersecretion is now being considered as a risk factor for increased morbidity. The irritant and epithelial membrane effects of O3, a main component of urban smog, upon the airway, and in particular on mucin-type secretory cells and/or interaction with epithelial physiology, have not been investigated vigorously, and at best only superficially, in vivo. We have recently demonstrated in genetically diverse inbred mice that O3-induced pulmonary inflammation and up-regulation of lung mucin secretion and airway mucociliary clearance are host factor dependent. These results match translationally with our evaluations in humans where O3 exposure leads to alterations in mucociliary clearance, and release of a mediator(s) capable of increasing mucin protein synthesis and secretion in vitro. Importantly additional observations by us in a healthy cohort of non-smoking human subjects (n=135) demonstrates that a homozygotic genotype for a single nucleotide polymorphism of the quinone oxido-reductase enzyme, NQO1, protects from the acute irritant effects on air flow that occur with exposure to ambient levels of O3. We have also found that NQO1 can modulate synthesis of mucin proteins by airway epithelial cells in vitro; and in connection with host-factor dependency, that NQO1 is differentially expressed in mice models susceptible and resistant to O3. As a working global hypothesis we propose that exposure to O3 by susceptible humans activates NQO1, generates reactive oxygen metabolites and leads to an increase in MUC5AC mRNA expression and production of mucins by airway epithelial cells. This cycle is re-initiated when O3-induced airway neutrophilia, leads to re-activation of NQO1 by neutrophil elastase, leading to expression and secretion of mucins, disordered mucociliary clearance, and reduced pulmonary function. Investigations are proposed for mice models represented by an O3 susceptible strain, a lung mucin hypersecretion model, and a NQO1 deficient model and simultaneous with translational studies in humans that are segregated genetically between wild-type (NQO1 sufficient) and a single nucleotide polymorphism associated with NQO1 deficiency. The research plan is the initial step towards a definitive link between an ubiquitous urban air pollutant, and genetic factors that regulate oxidant-induced airway hypersecretion of mucus.

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:subjects with current or past smoking history, acute respiratory illness within six weeks of the study, and significant non-pulmonary disease as determined by the investigator, pregnancy, age <18 or >35 yr, or inability to understand the protocol. Subjects will be requested to refrain from anti-histamines, nonsteroidal anti-inflammatory agents, and supplemental vitamins, e.g. C and E, for 1 week prior to, and during lab visits for exposures and follow-up measures.

-

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Subjects will be healthy adults, non-smokers, recruited from the University campus and local community. Fifty% will be female. Recruitment of minority ethnic groups will be consistent with census population for central NC. Subjects will have a clinical history and lung function screening at protocol entry. Female subjects of childbearing age will have pregnancy testing. Equal numbers of NQO1 sufficient and deficient subjects, based upon genoytypic pre-screening and stratified by racial background will be studied. Subjects will also be genotyped for GSTM1 wild type or null genotype. As individuals with an increased BMI may respond strongly to O3 we will only recruit subjects with body habitus within normal range for gender, age, and racial group.
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2008-08; Primary Completion 2011-10 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Airway Mucociliary Clearance | 6-24 h post-exposure to filatered air or ozone.

SECONDARY OUTCOMES:
Bronchial Epithelial Cells obtained by bronchoalveolar lavage. | 6-24 h post-exposure to filtered air or ozone.

CONTACTS AND LOCATIONS:
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States